CLINICAL TRIAL: NCT04283201
Title: Development, Implementation and Evaluation of the Effectiveness of Recommendations for the Prevention of Type 2 Diabetes in Ukraine
Brief Title: Type 2 Diabetes Mellitus Prevention Ukraine
Acronym: T2DPUA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Komisarenko Institute of Endocrinology and Metobolism (Other Government)
Responsible Party: Principal Investigator, Mykola Khalangot, Clinical Professor, Principal Investigator, Komisarenko Institute of Endocrinology and Metobolism
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0118U002166
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Impaired Fasting Glucose; Impaired Glucose Tolerance; Type 2 Diabetes
Keywords: lifestyle modification; type 2 diabetes; prevention; Ukraine; Rural
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 30 persons from this category were additionally advised to consume insoluble dietary fiber 15 g per day (Vitacel wheat fiber) for 3 months, after which a repeat anthropometric and biochemical study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet (Experimental)
  Interventions: Other: Macronutrient modification
- Physical activity (Experimental)
  Interventions: Other: Physical activity; Other: Macronutrient modification

INTERVENTIONS:
Other: Physical activity — Moderate activity 150 min per week
  Arms: Physical activity
Other: Macronutrient modification — Insoluble dietary fiber 15 g per day (Vitacel wheat fiber); sugar limitation

SUMMARY:
Development, implementation and evaluation of the effectiveness of lifestyle recommendations for the prevention of type 2 diabetes in rural population of Ukraine

DETAILED DESCRIPTION:
An oral glucose tolerance test and anthropometric measurements were performed for 300 randomly selected rural residents of the Kyiv region of Ukraine. Persons from impaired glucose regulation category (impaired fasting glucose - IFG) was enrolled to diabetes prevention intervention study (T2DPUA).

Individuals in the IFG category received advice on limiting sugar intake (not more than 25 g per day), increasing physical activity (30 minutes daily). 30 persons from this category were additionally advised to consume insoluble dietary fiber 15 g per day (Vitacel wheat fiber) for 3 months, after which a repeat anthropometric and biochemical study. Objective control of physical activity and body composition is also provided.

ELIGIBILITY:
Inclusion Criteria:

Persons with fasting blood glucose level >=6.1 mmol/l; persons aged 18-79 who signed an informed consent for the study.

Exclusion Criteria:

Known diabetes; acute infectious diseases; other serious diseases

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
New type 2 diabetes cases | 3 month
  fasting blood glucose level >=6.1 mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Victor Kravchenko, PhD, Prof, Study Director — V.P.Komisarenko Institute of Endocrinology and Metabolism
Locations (1):
- V.P.Komisarenko Institute of Endocrinology and Metabolism, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No